CLINICAL TRIAL: NCT01029613
Title: Adalimumab in Rheumatoid Arthritis. An Investigation of Changes in Disease Activity and Course of Joint Destruction by Use of 3 Tesla Whole-Body MRI, Dedicated 3 Tesla MRI and CT of the Hand, and Soluble Biomarkers
Brief Title: Adalimumab in Rheumatoid Arthritis. An Investigation of Wholebody MRI, Conventional MRI, CT and Circulating Biomarkers
Status: Completed | Type: Observational
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, MOstergaard, Professor, Glostrup University Hospital, Copenhagen
Other Study IDs: WRAP
Record Dates: First submitted 2009-12-09; First posted 2009-12-10 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Rheumatoid arthritis
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab — sc. inj. Humira 40 mg every other week from week 0 to 52

SUMMARY:
Adalimumab in rheumatoid arthritis. An investigation of changes in disease activity and course of joint destruction by use of 3 Tesla Whole-Body MRI, dedicated 3 Tesla MRI and CT of the hand, and soluble biomarkers. Furthermore to compare ultrasound examination with wholebody MRI etc.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old and < 85 years old
* RA in accordance with American College of Rheumatology 1987 criteria
* Moderate or highly active RA defined as DAS28 > 3,2 (CRP based)
* Clinical indication for TNF-α inhibitor treatment by the treating physician
* No contraindications for TNF-α inhibitor treatment
* No contraindications for MRI
* Serum creatinine in normal range
* Sufficient contraception for fertile women
* Capable of giving informed consent
* Capable of complying with the examination program of the protocol

Exclusion Criteria:

* Other DMARDs than MTX from less than 4 weeks before inclusion and throughout the study period
* Cyclophosphamide, Chlorambucil or other alkylating agents from less than 4 weeks before inclusion and throughout the study period
* Intramuscular or intravenous injection of glucocorticoid from less than 4 weeks before inclusion and throughout the study period
* Pregnancy wish, pregnancy or breast-feeding
* Contraindications for TNF-α inhibitor treatment
* Contraindications for MRI
* Known recent drug or alcohol abuse
* Failure to provide written consent
* Incapable of complying with the examination program for physical or mental reasons

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rheumatoid arthritis according to the ACR criteria (1987) with high disease activity starting TNF-alpha inhibitor
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2009-12; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
EULAR response criteria | 16 weeks

SECONDARY OUTCOMES:
Number of joints with inflammation on MRI | 16 and 52 weeks
Erosions on X-rays and CT | 52 weeks
Biomarkers | 16 and 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mikkel Østergaard, Professor, Principal Investigator — Dep. of Rheumatology, Glostrup Hospital; Susanne J Pedersen, MD, Study Chair — Dep. of Rheumatology, Glostrup Hospital
Locations (8):
- Denmark (8):
  - Dep. of medicine, Herlev Hospital, Copenhagen
  - Dep. of Radiology, Herlev Hospital, Copenhagen
  - Dep. of Rheumatology, Frederiksberg and Bispebjerg Hospitals, Copenhagen
  - Dep. of Rheumatology, Gentofte Hospital, Copenhagen
  - Dep. of Rheumatology, Glostrup Hospital, Copenhagen
  - Dep. of Rheumatologym Glostrup Hospital, Copenhagen
  - Dep. of Rheumatology, Helsingør Hospital, Hørsholm
  - Dep. of Rheumatology, Køge Hospital, Køge